CLINICAL TRIAL: NCT03709615
Title: Therapeutic Processes in Internet-Based CBT for Social Anxiety Disorder: A Randomized Controlled Trial.
Brief Title: Therapeutic Processes in iCBT for SAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Hebrew University of Jerusalem (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Idan Moshe Aderka, Principal Investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHaifaCBT
Record Dates: First submitted 2017-12-11; First posted 2018-10-17 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Social Anxiety Disorder; Social Phobia
Keywords: Social anxiety disorder; iCBT; Therapeutic processes
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait list (No Intervention): Wait list condition with no active treatment, length of 10 weeks, with weekly measurements.
- Intervention- active treatment (Experimental): Internet delivered CBT for social anxiety disorder
  Interventions: Behavioral: Internet delivered CBT for social anxiety disorder

INTERVENTIONS:
Behavioral: Internet delivered CBT for social anxiety disorder — An internet-based CBT for social anxiety based on a protocol from Andersson et al., 2006:
  "Internet-based self-help with therapist feedback and in vivo group exposure for social phobia: a randomized controlled trial."
  Arms: Intervention- active treatment

SUMMARY:
The current study examines therapeutic processes during internet-based cognitive-behavioral therapy for social anxiety disorder. Participants will be randomized to either treatment or wait-list conditions. Participants in the wait-list condition will receive active treatment following the wait-list period.

DETAILED DESCRIPTION:
Internet-based cognitive-behavioral therapy (iCBT) is an effective treatment for social anxiety disorder (SAD). However, little is known about the processes and mechanisms of change in this treatment. Compared to face to face (FTF) treatments, online interventions may operate through partially different mechanisms of change due to the text-based nature of the interaction and the reduced level of therapist involvement. The present randomized controlled trial will examine therapeutic processes during iCBT for SAD including the presence of sudden gains and their relationship to outcome, the relationship between anxiety and depressive symptoms along the course of treatment, changes in the therapeutic alliance and attrition from therapy. Moreover, we will compare iCBT for SAD with a wait-list control group and utilize weekly measurements of anxiety, depression, and SAD-related cognitions in both groups. This will facilitate comparison between temporal processes in both conditions and also shed light on processes occurring in wait-list conditions.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-5 criteria for social anxiety disorder.
* Fluency in Hebrew
* Access to internet

Exclusion Criteria:

* Substance use disorders
* Past or present psychosis
* High levels of suicidality
* Changes in pharmacological treatment 3 months or less prior to the start of the trial
* Participation in other psychotherapeutic treatments during the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Social anxiety severity | Change from Baseline LSAS at post treatment (12 weeks)
  Post treatment Liebowitz Social Anxiety Scale (LSAS). Score ranges from 0 to 144 where higher score indicates more sever social anxiety
Diagnosis of SAD based on clinical interview | Change from Baseline ADIS diagnosis at post treatment (12 weeks)
  Diagnoses derived from the Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS)
Social anxiety severity | Change from Baseline LSAS at 6 months follow-up
  Follow-up Liebowitz Social Anxiety Scale (LSAS). Score ranges from 0 to 144 where higher score indicates more sever social anxiety

SECONDARY OUTCOMES:
Social anxiety severity - additional measure | Change from Baseline SPIN at post treatment (12 weeks)
  Post treatment Social Phobia Inventory (SPIN). Score ranges from 0 to 68 where higher score indicates more sever social anxiety
Social anxiety severity - additional measure | Change from Baseline SPIN at 6 months follow-up
  Post treatment Social Phobia Inventory (SPIN). Score ranges from 0 to 68 where higher score indicates more sever social anxiety

OTHER OUTCOMES:
Depressive symptoms severity | Change from Baseline BDI-II at post treatment (12 weeks)
  Post treatment Beck Depression Inventory II, (BDI-II). Score ranges from 0 to 63 where higher score indicates more sever depression.
Depressive symptoms severity | Change from Baseline BDI-II at 6 months follow-up
  Post treatment Beck Depression Inventory II, (BDI-II). Score ranges from 0 to 63 where higher score indicates more sever depression.

CONTACTS AND LOCATIONS:
Overall Officials: Idan M Aderka, PhD, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shalom JG, Strauss AY, Huppert JD, Andersson G, Aderka IM. A theoretically based experimental manipulation of the processing of sudden gains: Considering reasons, meaning, and opportunities to leverage the gain. J Consult Clin Psychol. 2025 Feb;93(2):120-130. doi: 10.1037/ccp0000941. Epub 2024 Dec 30. PMID 39913487
- [Derived] Shalom JG, Strauss AY, Huppert JD, Andersson G, Agassi OD, Aderka IM. Predicting sudden gains before treatment begins: An examination of pretreatment intraindividual variability in symptoms. J Consult Clin Psychol. 2020 Sep;88(9):809-817. doi: 10.1037/ccp0000587. Epub 2020 Jun 25. PMID 32584117